CLINICAL TRIAL: NCT04143152
Title: Evaluation of a Biomarker Panel for the Diagnosis and Prognosis of Pancreatic Cancer
Brief Title: Pancreatic Cancer Biomarker Study
Status: Active, not recruiting | Type: Observational
Sponsor: Van Andel Research Institute (Other)
Collaborators: Corewell Health West (Other); Mercy Health (Other)
Responsible Party: Sponsor
Other Study IDs: 19021
Record Dates: First submitted 2019-10-16; First posted 2019-10-29 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diagnostic/prognostic cohort: Patients being evaluated for a potential pancreatic abnormality or for potential treatment for pancreatic adenocarcinoma.
- Surveillance Cohort: Patients who are being monitored for recurrence following surgical or medical treatment for pancreatic adenocarcinoma

SUMMARY:
This is a non-treatment, blood collection study to evaluate biomarker panels for the diagnosis and prognosis of pancreatic cancer.

DETAILED DESCRIPTION:
This is a non-treatment, blood collection study to evaluate biomarker panels for the diagnosis and prognosis of pancreatic cancer.

Study participants will be recruited by physician referral or from a list of clinical patients being evaluated for a potential pancreatic abnormality or for potential treatment of pancreatic cancer. Additionally, a surveillance cohort will be recruited among individuals who are being monitored for recurrence following surgical or medical treatment for pancreatic cancer.

Peripheral blood specimens will be collected from all participants at time of enrollment. Additional specimens may be collected from surveillance cohort participants no more frequently than once every 3 months as clinically indicated.

The specimens will be sent to a clinical lab for sTRA biomarker and CA19-9 analysis. Participants will be followed for 36 months to track clinical outcomes. The performance of the investigation biomarker for the diagnosis, prognosis, or surveillance of pancreatic cancer will be compared to the performance of CA19-9.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis/Prognosis Cohort

* Patients being evaluated for possible pancreatic abnormality, via additional radiological test (endoscopic ultrasound, abdominal CT scan), blood test (CA19-9), or other diagnostic procedure.
* Patients being evaluated for medical or surgical treatment for pancreatic cancer or pancreatitis on the basis of previous clinical and radiological findings.

Surveillance Cohort

* Patients being monitored or who will be monitored for potential recurrence of pancreatic cancer following surgical or medical treatment of pancreatic adenocarcinoma.

Exclusion Criteria:

* The participant is unwilling or unable to provide written informed consent.
* In the investigator's opinion, the participant is unsuitable for the study.
* The participant does not speak English.
* The participant is a prisoner.
* The participant is known to be pregnant.
* The participant is less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from collaborating clinical sites by screening physician schedules and through physician referral.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of adenocarcinoma of the pancreas | Up to three years
  Number of patients clinically diagnosed with pancreatic adenocarcinoma
Investigational biomarker panel for diagnosis | Enrollment
  sTRA biomarker and CA 19-9 levels at enrollment

SECONDARY OUTCOMES:
Disease progression | Up to three years
  Disease progression of pancreatic adenocarcinoma as measured by RESIST v1.1 criteria
Investigational biomarker panel for disease surveillance | Up to three years
  sTRA biomarker and CA 19-9 levels measured at any time point deemed clinically relevant for standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Haab, PhD, Principal Investigator — Van Andel Research Institute
Locations (1):
- Mercy Health Saint Mary's Hospital, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Staal B, Liu Y, Barnett D, Hsueh P, He Z, Gao C, Partyka K, Hurd MW, Singhi AD, Drake RR, Huang Y, Maitra A, Brand RE, Haab BB. The sTRA Plasma Biomarker: Blinded Validation of Improved Accuracy Over CA19-9 in Pancreatic Cancer Diagnosis. Clin Cancer Res. 2019 May 1;25(9):2745-2754. doi: 10.1158/1078-0432.CCR-18-3310. Epub 2019 Jan 7. PMID 30617132